CLINICAL TRIAL: NCT05156697
Title: The ACTivating Fat OXidation Through Capsinoids (ACTIFOX) Study
Brief Title: ACTivating Fat OXidation Through Capsinoids
Acronym: ACTIFOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Junta de Andalucia (Other Government); Spanish Ministry of Education (FPU16/02828, FPU16/05159) (Unknown); Spanish Ministry of Economy and Competitiveness (PTA 12264-I) (Unknown)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 839/CEIH/2019
Record Dates: First submitted 2021-11-12; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Overweight and Obesity
Keywords: capsinoids; dihydrocapsiate; FATmax; MFO; aerobic exercise; nutraceuticals; food ingredients
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo + Exercise (Placebo Comparator): Placebo pills + 60 min of aerobic exercise
  Interventions: Other: Placebo + Exercise
- Dihydrocapsiate + Exercise (Experimental): 12 mg of dihydrocapsiate pills + 60 min of aerobic exercise
  Interventions: Dietary Supplement: Capsinoids + Exercise

INTERVENTIONS:
Dietary Supplement: Capsinoids + Exercise — 60 minutes of aerobic exercise (cycle-ergometer) at FATmax intensity + supplementation with 12 mg of dihydrocapsiate (7 min before starting the aerobic exercise)
  Arms: Dihydrocapsiate + Exercise
Other: Placebo + Exercise — 60 minutes of aerobic exercise (cycle-ergometer) at FATmax intensity + placebo pills (7 min before starting the aerobic exercise)
  Arms: Placebo + Exercise

SUMMARY:
Prior evidence suggests that capsinoids ingestion may increase resting energy expenditure (EE) and fat oxidation (FATox) in humans, although whether they can modulate those parameters during exercise conditions remains poorly understood. Investigators aimed to determine the effects of dihydrocapsiate (DHC) ingestion on EE and FATox during an acute bout of aerobic exercise at FATmax intensity (the intensity that elicits maximal fat oxidation [MFO] during exercise) in overweight/obese men.

A total of 24 sedentary overweight/obese men participated in this randomized, triple-blinded, placebo-controlled, crossover trial. On the first day, participants underwent a submaximal exercise test in a cycloergometer to determine their MFO and FATmax intensity during exercise. After 72 hours had elapsed, the participants returned in 2 further days (≥ 72 hours apart) and performed a 60 min steady-state test (SST, i.e., cycling at their FATmax, constant intensity) after ingesting either 12 mg of DHC or placebo; these conditions were randomized. Respiratory gas exchange was monitored by indirect calorimetry. Serum markers concentrations (glucose, triglycerides, and non-esterified fatty acids), skin temperature, thermal perception, heart rate and perceived fatigue were assessed as secondary outcomes.

DETAILED DESCRIPTION:
The study protocol and design have been approved by the Human Research Ethics Committee of the University of Granada (n°839/CEIH/2019) and the Servicio Andaluz de Salud and adhered to the tenets of the Declaration of Helsinki as revised in 2013.

Participants were asked to confirm having commuted to the research center by car, bus, tram, or motorcycle, having slept, as usual, having refrained from stimulant beverages within 24 h, and having avoided any moderate or vigorous physical activity within 24 h and 48 h (respectively).

METHODS SUMMARY

Briefly, in the first visit, sociodemographic and lifestyle data were registered, and medical screening was performed, blood samples were collected, and anthropometry and body composition measures were taken. On the second visit, the MFO during exercise and cardiorespiratory fitness (peak volume of oxygen consumption, VO2 peak) were respectively assessed through a submaximal exercise test coupled to a maximal effort test. On visits third and fourth, participants performed a 60 min steady-state exercise bout on a cycle ergometer at FATmax intensity (i.e., at the intensity at which MFO is elicited) after having ingested either 12 mg of DHC or placebo. The conditions (DHC or placebo) on visits 3 and 4 were randomized. The washout period between visits 3 and 4 was ≥72 h. Of note, all exercise tests took place at a strictly controlled temperature of 22-23 ºC, given that environmental temperature largely influences EE and FATox.

EXTENDED METHODS

MEDICAL SCREENING, SOCIODEMOGRAPHIC DATA COLLECTION, AND ANTHROPOMETRY AND BODY COMPOSITION ASSESSMENTS:

On the first visit, participants arrived at the research center at 08:00 h, in fasting conditions (8 h). Participants were informed about the study protocols details and gave their oral and written informed consent to participate in the study. Sociodemographic data and data related to participants´ dietary habits (including pungent consumption), appetite, physical activity levels, sleep, and other lifestyle habits were recorded by questionnaires (some of them filled at home). Afterward, a medical doctor conducted an anamnesis to ensure that each participant was in suitable physical conditions to participate in the study and to practice exercise. Next, participants underwent an electrocardiogram in resting conditions, which was conducted by an expert medical doctor. Systolic and diastolic blood pressure were also measured with an automatic sphygmomanometer (Omron M2; Omron Healthcare, Kyoto, Japan). These measurements were repeated on 3 consecutive occasions and the average systolic and diastolic blood pressure were calculated. Only participants presenting a non-risk medical history and normal electrocardiogram were allowed to participate in the study. Blood samples were collected from the antecubital vein in the morning (8.00-9.00 am), with subjects sitting and in resting conditions. Blood samples were collected in serum Vacutainer Tubes® (Vacutainer® SST™ II Advance tubes) and centrifuged following the manufacturer's instructions. Afterward, serum samples were sent to the hospital lab for the analysis of the analytes of interest.

Anthropometry and body composition assessments also took place on the first visit. Body weight and height were measured (no shoes, light clothing) using a model 799 Seca scale and stadiometer (Seca, Hamburg, Germany). Waist circumference was measured twice at the minimum perimeter area with a measuring tape (mm precision), and the mean value was calculated. For those participants with abdominal obesity, waist circumference was measured just above the umbilicus (horizontal plane). Body fat mass and percentage, lean body mass, and visceral adipose tissue (VAT) mas were then measured by whole-body dual-energy X-ray absorptiometry (HOLOGIC, Discovery Wi, Marlborough, MA). Body mass, lean mass, and fat mass indexes were calculated as kg/m2.

SUBMAXIMAL AND MAXIMAL EXERCISE TESTS:

On the second visit, individuals arrived at the research center normally between 15:30 and 19:00. Participants confirmed having met the above-stated pre-experimental conditions, as well as arriving in fasting conditions (5-6 h) and having followed a standardized diet that participants were instructed to follow during the previous day. Then, participants urinated, dressed as above, and entered a quiet, warm (22-23 °C) room. A submaximal-graded exercise test was performed (to determine the MFO) coupled to a maximum effort test (used to determine the VO2peak) employing an Ergoselect 200 cycle ergometer (Ergoline GmbH, Lindenstrasse, Germany). More in detail, the submaximal exercise protocol coupled to indirect calorimetry started with a 3 min stage at 20 watts (W) as a warm-up, followed by increments of 20 W every 3 min, until resting exchange ratio (RER) was ≥1 at least for 30 s (as determined by indirect calorimetry). At this point, the maximal exercise protocol started (with no interruptions), and increments of 20 W took place every 1 min until volitional exhaustion was reached, or participants had to stop because of peripherical fatigue. Of note, the cycling power values (W) at which MFO happened for each individual were used as the target exercise intensity (i.e. FATmax) for the subsequent steady-state tests. Through the exercise test, participants' perceived fatigue was assessed using a rating of the reported perceived exertion (RPE) scale, and heart rate was measured using a Polar RS800 heart-rate monitor (Polar Electro Inc., Woodbury, NY, USA). Respiratory gas exchange was monitored with a CPX Ultima CardioO2 system (Medical Graphics Corp., St Paul, MN) with a facemask model 7400 (Hans Rudolph Inc., Kansas City, MO), and a preVent™ metabolic flow sensor (Medical Graphics Corp.). Oxygen consumption (VO2) was measured using a galvanic fuel cell and carbon dioxide production (VCO2) was assessed using a non-dispersive infrared sensor. According to the manufacturer's recommendations, the gas analyzer was calibrated using standard gas concentrations immediately before each test.

STEADY-STATE EXERCISE TESTS:

On the third visit (≥72 h after the second day), and again on the fourth visit (≥72 h later to avoid carry-out effects), participants came to the laboratory and underwent the steady-state tests after the ingestion of DHC or placebo, in a randomized order. Participants arrived at the same time as on the second visit and confirmed having met exactly the same pre-experimental conditions. Participants urinated, dressed in standard clothing, and entered a quiet, warm (22-23 °C) room. A Polar RS800 heart-rate monitor was placed on their chest using a chest wrap band. Then, a set of 16 DS-1922 L Button TM wireless thermometers (Thermochron, Dallas, TX, USA) were attached to the subject's skin in different places to monitor skin temperature changes through the experiment. They were put on the forehead, left pectoralis, left elbow region, left index fingertip, left forearm, rear neck central area, right clavicula, right deltoid, right shinbone, right sub-clavicular area, right supra-clavicular area, right thigh, and upper breastbone. Afterward, participants sat and stay relaxed for 10 min (resting period, timepoint -20´), and were instructed not to move nor cross their arms and legs, and their baseline skin temperature and heart rate measures were taken. The first intravenous blood sample was collected 10 min before starting the steady-state test (timepoint -10'). Immediately 3 min after the first blood collection (timepoint -7'), participants ingested either 12 mg of DHC (4 pills 3 mg each one) or placebo. Then participants sat in the cycle ergometer where the steady-state tests would be performed, and a gas mask was put on for the gases exchange measurement. The same metabolic cart as on the second visit was used. The gas collection started 1 min before the beginning of the steady-state test (timepoint -1') with the participants sitting in the cycle ergometer without pedaling. After 1 min of gases recording in resting conditions, the steady-state test at FATmax intensity started and continued until min 60, the moment at which the test was ended. Gases exchange and heart rate were continuously monitored. At time points 15', 30', 45', and 60', blood samples were collected.

TEST SUBSTANCES: DIHYDROCAPSIATE AND PLACEBO:

Investigators employed Capsiate Gold™ soft-gel capsules from Ajinomoto®. These capsules consisted of 3 mg of purified DHC vehiculated with canola oil, modified corn starch, vegetable glycerin, carrageenan, water, disodium hydrogen phosphate, and soy lecithin. Hemicellulose powder was used as a placebo. Both DHC and hemicellulose were encapsulated by independent manufacturers and put in different containers by an independent researcher (not involved in the current study). Each container was labeled with a different code (0 or 1) so that evaluators were not aware of the administered substance - therefore preventing bias. Of note, both DHC and placebo capsules looked exactly similar to unable the identification of the content by either researchers or participants.

ELIGIBILITY:
Inclusion Criteria:

* to be male
* to be 18-55 years old
* to be sedentary (<20 min moderate-to-vigorous physical activity on <3 days/week)
* to be non-smoker
* not to be under medication
* to have a stable body weight over the preceding three months (<3 kg change)

Exclusion Criteria:

* having been diagnosed with diabetes, hypertension, or any medical condition(s) that can interfere with or be aggravated by exercise
* using medication that could affect energy metabolism
* present a family history of CVD
* to have an abnormal electrocardiogram, regular and high consumption of spicy foods
* being frequently exposed to cold temperatures (e.g., indoors/outdoors workspace with low-temperatures, such as cold-storage works, ski/snow monitors, fieldworks during the winter sessions or low-temperatures areas)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in energy expenditure (kcal/day) by indirect calorimetry (CPX Ultima CardioO2 system) | It will be continuously measured through the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in fat oxidation (g/min) by indirect calorimetry (CPX Ultima CardioO2 system) | It will be continuously measured through the 60 minutes-bout of aerobic exercise at FATmax intensity

SECONDARY OUTCOMES:
Change in serum levels of glucose (mg/dL) by automated analyzer (Beckman Coulter) | It will be measured at timepoints 0, 15, 30, 45 and 60 minutes, of the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in serum levels of triglycerides (mg/dL) by automated analyzer (Beckman Coulter) | It will be measured at timepoints 0, 15, 30, 45 and 60 minutes, of the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in serum levels of non-esterified fatty acids (mmol/L) by automated analyzer (Beckman Coulter) | It will be measured at timepoints 0, 15, 30, 45 and 60 minutes, of the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in skin temperature (ºC) by iButtons wireless thermometers | It will be continuously measured through the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in thermal perception (unitless) by ASHRAE scales | It will be measured every 15 minutes of the 60 minutes-bout of aerobic exercise at FATmax intensity
Change in rated perceived exertion (unitless) by RPE scales | It will be measured every 5 minutes of the 60 minutes-bout of aerobic exercise at FATmax intensity

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Instituto Mixto Universitario Deporte y Salud - iMUDS, Granada
  - Instituto Mixto Universitario Deporte y Salud, Granada

REFERENCES:
- [Derived] Osuna-Prieto FJ, Acosta FM, Perez de Arrilucea Le Floc'h UA, Riquelme-Gallego B, Merchan-Ramirez E, Xu H, De La Cruz-Marquez JC, Amaro-Gahete FJ, Llamas-Elvira JA, Trivino-Ibanez EM, Segura-Carretero A, Ruiz JR. Dihydrocapsiate does not increase energy expenditure nor fat oxidation during aerobic exercise in men with overweight/obesity: a randomized, triple-blinded, placebo-controlled, crossover trial. J Int Soc Sports Nutr. 2022 Jul 19;19(1):417-436. doi: 10.1080/15502783.2022.2099757. eCollection 2022. PMID 35875695